CLINICAL TRIAL: NCT04084535
Title: Effects of Inspiratory Muscle Training vs. High Intensity Interval Training Program on the Recovery Capacity After a Maximal Dynamic Apnea in Breath-hold Divers. A Randomized Crossover Trial
Brief Title: Effects of High Intensity Interval Training (HIIT) vs. Inspiratory Muscle Training on the Recovery After a Maximal Apnea.
Acronym: (HIIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Fran de Asís Fernández, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS - PI - 215/2018
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Exercise Training; Respiratory Muscle Training; High-Intensity Interval Training; Apnea
MeSH Terms: conditions — Apnea | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Intervention Model: Crossover Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Active Comparator): It will apply a HIIT program for 4 weeks, with 3 sessions per week of 30 min per session, including warm-up, recovery between intervals and return to calm.
  Interventions: Other: High intensity interval training
- Inspiratory muscle training (Active Comparator): It will apply an inspiratory muscle training for 4 weeks, with 3 sessions per week of 30 min per session, including warm-up, recovery between intervals and return to calm.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: High intensity interval training — Participants will perform 3 HIIT sessions per week, involving 10 min of intense exercise within a time commitment of 30 min per session, including warm-up, recovery between intervals and cool down.
  Arms: High intensity interval training
Other: Inspiratory muscle training — Participants will perform 3 inspiratory resistance training sessions per week, involving 30 min per session, including warm-up, recovery between intervals
  Arms: Inspiratory muscle training

SUMMARY:
The aim of this randomized cross-over controlled study was to assess the effects of an 4-week exercise program on the recovery capacity after a voluntary maximal apnea. Participants will be randomly allocated to receive either a high intensity interval training (HIIT), or an inspiratory muscle training (IMT) using an inspiratory resistance device.

DETAILED DESCRIPTION:
It is a multi-center study. 3 different Spanish Freedivers Centres are included in the study (Madrid, Zaragoza, and Barcelona).

For each participant, exercise program started with one or the other program. Hence, both interventions were applied once with the participant randomly allocated to receive the same intervention. The trial included four study visits. Each exercise training program will be applied sessions per week during 4 weeks. Participants received baseline assessments at the beginning of nay intervention, and post-intervention assessments at the end of the fourth week. The wash-out period will be two weeks. After these two weeks participants switched intervention.

ELIGIBILITY:
Inclusion Criteria:

* Absence of pain or illness
* No changes in cognitive ability
* Over 18 years old.
* Member of the Spanish Federation of Underwater Activities.
* Positive medical examination that allows the diver to practice voluntary apnea.

Exclusion Criteria:

* People with systemic diseases, tumors, infections, pacemakers, history of epilepsy, hydrophobia, pregnancy women, pharmacological treatment.
* To be participating in other physical activities during the experimental research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation recovery | Before and after training intervention (after 4 weeks)
  Oxygen Saturation recovery will be record by the experimenters every 5 seconds by a handheld pulse-oximeter during the 1 min recovery time after a maximal dynamic apnea. The outcome represents the time it takes to get a 95% of saturation during these 1 minute.

SECONDARY OUTCOMES:
Lung function (forced spirometry) | Before and after training intervention (after 4 weeks)
  The Spirometry will be perform according to American Thoracic Society criteria and was measured in litres. The maneuver will be perform 3 times and recording the best one.
Maximum Respiratory Pressures | Before and after training intervention (after 4 weeks)
  The maximum respiratory pressures (MIP and MEP) will be measure with a device. This device applies an inspiratory/expiratory load which provides a resistance. The maneuver will be perform in a sitting position. Measuring a minimum of 3 times will be perform, recording the highest value.
Lactic acid recovery | Before and after training intervention (after 4 weeks)
  The level of lactic acid in the blood will be measure by a device that used a blood lactic acid measurement that you've gotten by the finger-stick method. It will be record by the experimenters 3 times: immediately after the maximal dynamic apnea, after 3 min and after 10 min of the maximal dynamic apnea.
Heart Rate recovery | Before and after training intervention (after 4 weeks)
  Heart Rate will be record by the experimenters every 5 seconds by a handheld pulse-oximeter during the 1 min recovery time after a maximal dynamic apnea. The outcome represents how long does it take before the participant periodic Heart Rate is stabilized during these 1 minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Madrid FREEDIVERS association, Madrid, Spain

REFERENCES:
- [Background] Andersson JP, Liner MH, Runow E, Schagatay EK. Diving response and arterial oxygen saturation during apnea and exercise in breath-hold divers. J Appl Physiol (1985). 2002 Sep;93(3):882-6. doi: 10.1152/japplphysiol.00863.2001. PMID 12183481